CLINICAL TRIAL: NCT06097377
Title: Lymphatic Magnetic Resonance Imaging Abnormalities in Children With Tetralogy of Fallot: A Case-Control Study
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Vibeke Brix Christensen, MD, DMSc, Rigshospitalet, Denmark
Other Study IDs: Lymphatic Magnetic Resonance
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Tetralogy of Fallot; Lymphatic
MeSH Terms: conditions — Tetralogy of Fallot

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ToF
- Controls

SUMMARY:
This study examines subclinical lymphatic abnormalities in Tetralogy of Fallot patients, utilizing lymphatic magnetic resonance and near-infrared fluorescence imaging.

ELIGIBILITY:
Inclusion Criteria:

* ToF

Exclusion Criteria:

-

Ages: 6 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: controls and ToF patients between 6 - 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Lymphatic abnormalities | During scan
  MRI assessed lymphatic abnormalities

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, København Ø, Denmark

IPD SHARING:
Plan to Share IPD: Undecided